CLINICAL TRIAL: NCT04310176
Title: Randomized Phase 2 Study of Valproic Acid in Combination With Bevacizumab and Oxaliplatin/Fluoropyrimidine Regimens in Patients With Ras-mutated Metastatic Colorectal Cancer
Brief Title: Valproic Acid in Combination With Bevacizumab and Oxaliplatin/Fluoropyrimidine Regimens in Patients With Ras-mutated Metastatic Colorectal Cancer
Acronym: REVOLUTION
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REVOLUTION; 2018-001414-15 (EudraCT Number)
Record Dates: First submitted 2019-11-25; First posted 2020-03-17 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-03

CONDITIONS: Ras-mutated Metastatic Colorectal Cancer
Keywords: Metastatic colorectal cancer; Ras mutations; Valproic acid
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Valproic Acid; Capecitabine; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (Active Comparator): Chemotherapy (mFOLFOX-6/mOXELL) + Bevacizumab for 12 cycles (24 weeks)
  Maintenance treatment (Standard): Fluoropyrimidines (5-Fluorouracil/Capecitabine) + Bevacizumab until disease progression or unacceptable toxicity
  Interventions: Drug: Bevacizumab; Drug: mFOLFOX6 regimen; Drug: mOXXEL regimen; Drug: Capecitabine; Drug: 5-fluorouracil
- Experimental (Experimental): Chemotherapy (mFOLFOX-6/mOXELL) + Bevacizumab + Valproic Acid administered oral daily from day -14 increasing doses and an intra-patient titration for a target serum level of 50-100µg/ml for 12 cycles (24 weeks)
  Maintenance treatment (Experimental): Fluoropyrimidines (5-Fluorouracil/Capecitabine) + Bevacizumab + Valproic Acid until disease progression or unacceptable toxicity
  Interventions: Drug: Bevacizumab; Drug: mFOLFOX6 regimen; Drug: mOXXEL regimen; Drug: Valproic acid; Drug: Capecitabine; Drug: 5-fluorouracil

INTERVENTIONS:
Drug: Bevacizumab — 5 mg/m2 as 20-to-30 minute intravenous (i.v.) infusion every two weeks. Maintenance treatment (both arms): 5 mg/m2 every 2 weeks (in combination with 5-Fluorouracil) or 7.5 mg/m2 every 3 weeks (in combination with capecitabine)
Drug: mFOLFOX6 regimen — Oxaliplatin 85 mg/m2 as 2-3 hours i.v. infusion on day 1 followed by levo-folinic acid 200 mg/m2 as 1- 2 hours i.v. infusion followed by i.v bolus. 5-fluorouracil 400 mg/m2, and a 46-hour i.v. infusion of 5-fluorouracil 2400 mg/m2 every two week
Drug: mOXXEL regimen — Oxaliplatin 85 mg/m2 as 2-3 hours i.v. infusion on day 1 plus oral capecitabine 1000 mg/m2 twice daily on days 1 to 10, every 2 weeks
Drug: Valproic acid — given orally from 500mg-1500mg daily and an intra-patient titration for a target serum level of 50-100µg/ml
  Arms: Experimental
Drug: Capecitabine — Maintenance treatment (both arms): 1250 mg/m2 twice daily on days 1 to 14, every 3 weeks or 1250 mg/m2 twice daily on days 1 to 10, every 2 weeks
Drug: 5-fluorouracil — Maintenance treatment (both arms): Levo-folinic acid 200 mg/m2 as 1- 2 hours i.v. infusion followed by i.v bolus. 5-fluorouracil 400 mg/m2, and a 46-hour i.v. infusion of 5-fluorouracil 2400 mg/m2 every two weeks

SUMMARY:
The primary aim of this study is to test whether the combination of valproic acid with bevacizumab and oxaliplatin/fluoropyrimidine regimens (mFOLFOX6/mOXXEL) can prolong progression free survival (PFS) as compared with bevacizumab and oxaliplatin/fluoropyrimidine regimens alone as first-line treatment in patients with metastatic colorectal cancer with mutation of RAS.

DETAILED DESCRIPTION:
Patients will be randomized 1:1 to receive oxaliplatin based chemotherapy (mFOLFOX6/mOXELL) plus bevacizumab for 12 cycles or the same chemotherapy plus bevacizumab and valproic acid for 12 cycle.

Thereafter, in both arms, patients who are progression free after 12 cycles (24 weeks) of treatment continue maintenance bevacizumab+fluoropyrimidines until disease progression or unacceptable toxicity.

Surgery may be carried out in case of appropriate tumour reduction is evident at response evaluation. Resectability has to be evaluated by a multidisciplinary review team and the decision regarding post-surgery chemotherapy is at the discretion of the investigators, according to the policy commonly adopted by their Institution in clinical practice.

ELIGIBILITY:
Inclusion criteria

* Age >=18 years
* Histologically confirmed diagnosis of colorectal adenocarcinoma
* Stage IV of disease (according to TNM 8th edition)
* RAS mutations
* Clinical or radiologic evidence of disease (at least one target or non target lesion according to RECIST 1.1)
* ECOG performance status 0 to 1
* Life expectancy > 3 months
* Use of an acceptable mean of contraception for men and women of childbearing potential
* Adequate recovery from previous surgery. At least 28 days should elapse from a surgical procedure or from performing a biopsy for the enrolment into the study
* Written informed consent

Exclusion criteria Cancer related

* RAS wild type colorectal cancer Prior, current or planned treatment related
* Prior chemotherapy or any other medical treatment for advanced colorectal cancer (previous adjuvant chemotherapy is allowed if ended > 6 months before relapse or > 24 months if the adjuvant treatment included oxaliplatin)
* Radiotherapy to any site for any reason within 28 days prior to randomization (palliative radiotherapy to bone lesions is allowed if >=14 days before randomization)
* Patient who have had prior treatment with an HDAC inhibitor and patients who have received compounds with HDAC inhibitor like activity, such as valproic acid
* Full dose anticoagulation with warfarin
* Current or recent (within the last 10 days) use of aspirin (>325 mg/day) or chronic use of other full dose nonsteroidal antiinflammatory drugs (NSAIDs) with antiplatelet activity Laboratory related
* Inadequate coagulation parameters:

  * activated partial thromboplastin time (APTT) >1.5 x or the upper limit of normal (ULN) or
  * INR >1.5
* Inadequate liver function, defined as:

  * AST/SGOT or ALT/SGPT >2.5 x ULN e/o serum (total) bilirubin >1.5 xULN for the institution
  * AST/SGOT or ALT/SGPT >5 x ULN e/o serum (total) bilirubin > 3 xULN for the institution in case of liver metastases.
* Inadequate renal function, defined as:

  * Creatinine clearance < 50 mL/min or serum creatinine >1.5 x ULN for the institution
  * urine dipstick for proteinuria >2pos. Patients with 1pos proteinuria at baseline dipstick analysis should undergo a 24hour urine collection and must demonstrate <=1g of protein in their 24hour urine collection
* Inadequate bone marrow function, defined as:

  * Neutrophils < 2000/mm3
  * Platelets < 100.000/ mm3
  * Hemoglobin (Hgb) < 9 g/dL Prior or concomitant conditions or procedures related
* Known dihydropyrimidine dehydrogenase (DPD) deficiency
* Pregnancy or breastfeeding
* Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure >100 mmHg on antihypertensive medications)
* History of any of the following within 6 months prior to randomisation: serious systemic disease, unstable angina, New York Heart Association (NYHA) Grade 2 or greater Congestive Heart Failure (CHF), clinically significant peripheral vascular disease, abdominal fistula, gastrointestinal perforation, or intra abdominal abscess
* History of arrhythmia, bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation which is symptomatic or requires treatment (CTCAE grade 3) or asymptomatic sustained ventricular tachycardia.
* Patients with long QT syndrome or QTc interval duration > 480 msec or concomitant medication with drugs prolonging QTc (see list in the appendix)
* Serious, non healing wound, ulcer, or bone fracture
* History of inflammatory bowel disease or active disease
* Evidence of bleeding diathesis or coagulopathy or other serious or acute internal bleeding within 6 months prior to randomization
* Central Nervous System (CNS) bleeding; history or clinical evidence of CNS stroke (hemorrhagic or thrombotic) within the last 6 months
* Inpatient surgical procedure, or significant traumatic injury within 28 days prior to randomization
* Minor surgical procedure, fine needle aspirations or core biopsy within 7 days prior to randomization
* Inability to take oral medication or requirement for intravenous (IV) alimentation or total parenteral nutrition with lipids, or prior surgical procedures affecting absorption
* Evidence of confusion or disorientation, or history of major psychiatric illness that may impair the patient's understanding of the Informed Consent Form or their ability to comply with study requirements
* Any other invasive malignancies within 5 years (except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer or surgically resected prostate cancer with normal PSA)
* Brain metastasis
* HIV positive patients
* Any other concomitant pathologies or laboratory alterations that prevent or contraindicate the use of study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-05-24 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | until progression of disease (up to 5 years)
  PFS is defined as the time elapsed from the date of randomization to the date of progression, as defined by investigators, or the date of death, whichever comes first

SECONDARY OUTCOMES:
centrally reviewed PFS (CR-PFS) | at week 12th and 24th and thereafter every 12 weeks until progression of disease (up to 5 years(
  FSCR is also measured as the time elapsed from the date of randomization to the date of progression, as defined by independent blind central review, or the date of death, whichever comes first
overall survival (OS) | 5 years
  OS is defined as the time elapsed from randomization to death due to any cause
Determination of changes in quality of life | at baseline, at week 12th and 24th and every 12 weeks thereafter until progression disease (up to 5 years)
  EORTC QLQ-C30, a quality of life questionnaires, composed by 30 items graded from1 (not at all) to 4 (very much) after 1 year from the diagnosis
Response rate | at week 12th and 24th and thereafter every 12 weeks until progression of disease (up to 5 years)
  according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Number of participants with treatment-related side effects | baseline, day 1 of each cycle and on maintenance treatment until progression disease (up to 5 years)
  graded according to Common Criteria for Adverse Events (CTCAE) version 5.0
metastases resection rate (R0/R1/R2) | up to 24 weeks
  determined at surgery (resection status) by pathologist follow: R0 no cancer cells at the resection margin; R1 microscopic positive margin, R2 macroscopic positive margin

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Avallone, MD, Principal Investigator — National Cancer Institute, Napoli; Maria Carmela Piccirillo, MD, Study Chair — National Cancer Institute, Napoli; Alfredo Budillon, MD, Study Chair — National Cancer Institute, Napoli
Locations (1):
- Istituto Tumori di Napoli - Fondazione G. Pascale, Napoli, Campania, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Avallone A, Piccirillo MC, Di Gennaro E, Romano C, Calabrese F, Roca MS, Tatangelo F, Granata V, Cassata A, Cavalcanti E, Maurea N, Maiolino P, Silvestro L, De Stefano A, Giuliani F, Rosati G, Tamburini E, Aprea P, Vicario V, Nappi A, Vitagliano C, Casaretti R, Leone A, Petrillo A, Botti G, Delrio P, Izzo F, Perrone F, Budillon A. Randomized phase II study of valproic acid in combination with bevacizumab and oxaliplatin/fluoropyrimidine regimens in patients with RAS-mutated metastatic colorectal cancer: the REVOLUTION study protocol. Ther Adv Med Oncol. 2020 Aug 11;12:1758835920929589. doi: 10.1177/1758835920929589. eCollection 2020. PMID 32849914
- See also: sponsor web-site for study conduction — https://usc.istitutotumori.na.it/